CLINICAL TRIAL: NCT05122169
Title: Establishment of Clinical Practice Guideline to Prevent Puerperal / Perinatal Infection in Vaginal Delivery for Pregnant Women and Newborns
Brief Title: Skip Prep of Vaginal Delivery to Prevent Puerperal / Perinatal Infection in Vaginal Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joong Shin Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Vaginal Delivery Skin Prep
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Vaginal Delivery; Surgical Site Infection
Keywords: Chlorhexidine-alcohol; Povidone-iodine; Perineal infection; Surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chlorhexidine (Experimental): Pre-vaginal delivery skip prep using chlorhexidine-alcohol
  Interventions: Drug: Chlorhexidine
- Povidone-iodine (Active Comparator): Pre-vaginal delivery skip prep using Povidone-iodine
  Interventions: Drug: Povidone-Iodine

INTERVENTIONS:
Drug: Povidone-Iodine — Skin preparation with povidone-iodine pre-vaginal delivery skin preparation.
  Other Names: Povidone-iodine 10%
  Arms: Povidone-iodine
Drug: Chlorhexidine — Skin preparation with chlorhexidine-alcohol pre-vaginal delivery skin preparation.
  Other Names: Hexitanol 2% Soln., Chlorhexidine Gluconate Solution
  Arms: chlorhexidine

SUMMARY:
This is a multi-center, randomized, controlled trial study to find whether use of chlorhexidine-alcohol or povidone-iodine for pre-vaginal delivery skin prep is superior to reduce postpartum infection in pregnant women with vaginal delivery. The primary outcome is the episiotomy site infection.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy
* Women who will undergo vaginal delivery after 37+0/7 weeks of gestation

Exclusion Criteria:

* Women who are allergy to chlorhexidine, alcohol, iodine, or shellfish
* Women with any infection at perineum (before vaginal delivery)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4140 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participant with episiotomy site infection | 21 days
  Superficial or deep infection of episiotomy site

REFERENCES:
- [Derived] Jung YM, Lee SM, Kim SY, Chung JH, Won HS, Lee KA, Park MH, Cho GJ, Oh MJ, Choi ES, Ahn KH, Hong SC, Sung JH, Roh CR, Kim SM, Kim BJ, Kim HJ, Oh KJ, Hong S, Park IY, Park JS. The Skin Antiseptic agents at Vaginal dElivery (SAVE) trial: study protocol for a randomized controlled trial. Trials. 2023 Feb 21;24(1):130. doi: 10.1186/s13063-023-07101-w. PMID 36810189